CLINICAL TRIAL: NCT01862913
Title: Computer-Assisted Cognitive-Behavioral Therapy for Adolescent Depression in Primary Care Clinics in Santiago, Chile (YPSA-M): A Randomized Controlled Trial
Brief Title: Computer-Assisted Cognitive-Behavioral Therapy for Adolescent Depression
Acronym: YPSA-M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Vania Martínez-Nahuel, Dr.med., University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FONDECYT Nº11121637
Record Dates: First submitted 2013-05-20; First posted 2013-05-27 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Depression
Keywords: depression; adolescents
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer-assisted CBT (Experimental): * Usual medical treatment in accordance with a decision algorithm based on the "Clinical Guidelines for the Treatment of Depression of the Ministry of Health of Chile".
  * Eight sessions of a computer-assisted cognitive-behavioral therapy. Trained psychologists administer this program in face to face meetings.
  Interventions: Other: Computer-assisted cognitive-behavioral therapy
- Usual care treatment (Active Comparator): - Usual psychological and medical treatment in accordance with a decision algorithm based on the "Clinical Guidelines for the Treatment of Depression of the Ministry of Health of Chile".
  Interventions: Other: Usual care treatment

INTERVENTIONS:
Other: Computer-assisted cognitive-behavioral therapy — The intervention arm will receive eight sessions of computer-assisted CBT plus usual medical treatment, as described in the AUGE Clinical Guidelines for Depression. Computer-assisted CBT sessions will be delivered on a weekly basis and assisted by trained psychologists in face-to-face meetings. The program is called 'Yo pienso, siento y actúo mejor' (YPSA-M); in English, 'I think, feel, and behave better'. Topics covered in the program will include information on symptoms and causes of depression, treatment options, problem-solving techniques and other cognitive-orientated strategies to challenge negative thoughts.
  Arms: Computer-assisted CBT
Other: Usual care treatment — The control arm will receive treatment as usual from the primary care clinics. The professionals in the primary care centers will be instructed to follow the AUGE Clinical Guidelines for Depression.
  Arms: Usual care treatment

SUMMARY:
Background: Most adolescents suffering depression are treated in primary care clinics. Cognitive-behavior therapy (CBT) is effective in the treatment of adolescent depression. The availability of appropriately trained CBT therapist may be limited, especially in primary care clinics. One way to increase the availability of CBT is to use computer-assisted CBT (c-CBT). It can be effective in the treatment of adults, although the outcomes in adolescents remain unclear.

Purpose: The purpose of this study is to determine whether a computer-assisted cognitive-behavioral therapy is effective for the treatment of depression in adolescents between 15 and 19 years of age in 4 primary care clinics in Santiago, Chile.

Study design: A two-arm single-blind (outcomes assessor) randomized controlled trial will be carried out with 216 adolescents. The efficacy, the adherence, and acceptability of the computerized-assisted cognitive behavioral therapy will be evaluated.

DETAILED DESCRIPTION:
This is a two-arm, single-blind (blinded only to outcome assessor), individually randomized controlled trial, which will compare the efficacy of computer-assisted CBT versus usual treatment for depression in adolescents in primary care clinics in Santiago, Chile.

General aim To carry out a randomized controlled trial to compare the efficacy of a computer-assisted CBT intervention versus usual care to treat depression in adolescents in primary care clinics in Santiago, Chile.

Specific aims

1. To compare the level of depressive symptoms of adolescents suffering depression treated with computer-assisted CBT versus usual care in primary care clinics.
2. To compare the level of dysfunctional thoughts, strategies for solving problems, and health-related quality of life (HRQoL) of adolescents suffering depression treated with computer-assisted CBT versus usual care in primary care clinics.
3. To compare adolescents' adherence to computer-assisted CBT versus usual care in primary care clinics.
4. To compare adolescents' satisfaction with computer-assisted CBT versus usual care in primary care clinics.

Hypotheses

1. Adolescents receiving the intervention will achieve lower scores (difference in mean of at least 0.4 standard deviations) in the depression questionnaire than those receiving the usual care, four months after randomization.
2. Adolescents receiving the intervention would have fewer dysfunctional thoughts than those receiving the usual care, four months after randomization.
3. Adolescents receiving the intervention would be better at solving problems than those receiving the usual care, four months after randomization.
4. Adolescents receiving the intervention would have better HRQoL than those receiving the usual care, four months after randomization.
5. Symptomatic improvements achieved at four months after randomization will be maintained at six months after randomization.

Setting and population Adolescents between 15 and 19 years of age attending four primary care clinics located in Puente Alto, a low-income municipality of Santiago, Chile, with a large adolescent population.

Training of primary care center professionals Before the start of recruitment, professionals in the four participating primary care centers will receive a special training session from the principal investigator to assist with the correct identification, diagnosis, and treatment of patients with depression, according to the AUGE Clinical Guidelines for Depression. There will also be a refresher session 6 months after the start of recruitment.

Recruitment Adolescents eligible for the study will be identified by health professionals of the four primary care clinics, as well as by psychologists and counselors of nearby schools, who will be informed of the study, trained to identify potential cases of depression among their students, and instructed to refer any adolescent who seems to have depression symptoms to the primary care clinics for further evaluation and possible participation in the study, according to inclusion and exclusion criteria.

Group assignment Those adolescents who at baseline assessment meet the inclusion criteria and do not meet the exclusion criteria will be randomly assigned to the intervention arm or to the control arm. Blocked (size of four), stratified randomization will be used. Stratification will be implemented regarding sex and severity of depression (mild, moderate, and severe) according to BDI score. Randomization will be generated using web-based random allocation algorithms. Allocation concealment will be carried out by keeping treatment assignment in numbered sealed envelopes in a central place; the envelopes will be opened by individuals who do not participate in the recruitment process.

Data collection All participants will be assessed at baseline and at four and six months after randomization. The instruments that will be used are all self-report questionnaires, which will be completed on paper by the participants. Trained psychologists who are blind to the group assignments will be present to assist the adolescents if necessary.

Data management After the participants have completed the questionnaires, the data will entered into a secure platform, without identifying information (each participant will be assigned an ID number). The original copies of the instruments will be filed and stored, under lock and key, in the principal investigator's office, along with the list linking the participants' names and ID numbers. Only two research assistants, in charge of data entry, and the statistician will have access to the database.

Data analysis Data and presentation of the results will be in accordance with CONSORT guidelines for randomized clinical trials, with the primary comparative analysis being conducted on an intention-to-treat basis. Initially, we will conduct descriptive analysis to assess the balance between the two groups. The primary analysis will employ multivariable linear regression to investigate differences in mean symptom scores (primary outcome measure) between groups at four months after randomization, adjusting for baseline outcome variable if imbalances are identified. Sensitivity analysis making different assumptions will be conducted to investigate the potential effects of missing data. Similar analyses will be conducted for the secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Beck Depression Inventory > o = 10
* Meets diagnostic criteria of a depressive disorder according Kiddie Sads Present and Lifetime Version interview (K-SADS-PL)
* Parent or caregiver giving informed consent and adolescent giving informed assent

Exclusion Criteria:

* Suicidal risk requiring in-patient care
* Bipolar Disorder
* Current substance dependence
* Current alcohol dependence
* Current psychosis
* Low intellectual abilities
* Current treatment with antidepressant and/or psychotherapy

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 216 (Actual)
Dates: Start 2013-06; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Beck Depression Inventory (BDI) at 4 months | Baseline and 4 months

SECONDARY OUTCOMES:
Change from baseline in Children's Automatic Thought Questionnaire (CATS) | Baseline, 4 months, and 6 months
Change from baseline in Social Problem Solving Inventory-Revised Short Form (SPSI-RS) | Baseline, 4 months, and 6 months
Change from baseline in KIDSCREEN-27 | Baseline, 4 months, and 6 months
  Health-related quality of life questionnaire
Change from baseline in Beck Depression Inventory (BDI) at 6 months | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vania Martínez-Nahuel, Dr.med., Principal Investigator — University of Chile
Locations (1):
- CESFAM Bernardo Leighton, CESFAM Cardenal Raúl Silva Henríquez, CESFAM Padre Manuel Villaseca, CESFAM San Gerónimo, Santiago, Chile

REFERENCES:
- [Derived] Martinez V, Rojas G, Martinez P, Gaete J, Zitko P, Vohringer PA, Araya R. Computer-Assisted Cognitive-Behavioral Therapy to Treat Adolescents With Depression in Primary Health Care Centers in Santiago, Chile: A Randomized Controlled Trial. Front Psychiatry. 2019 Jul 30;10:552. doi: 10.3389/fpsyt.2019.00552. eCollection 2019. PMID 31417440
- [Derived] Martinez V, Martinez P, Vohringer PA, Araya R, Rojas G. Computer-assisted cognitive-behavioral therapy for adolescent depression in primary care clinics in Santiago, Chile (YPSA-M): study protocol for a randomized controlled trial. Trials. 2014 Aug 5;15:309. doi: 10.1186/1745-6215-15-309. PMID 25091593